CLINICAL TRIAL: NCT03835169
Title: Intra Hospital Mortality Risk Factors in Patients Admitted to Cardiac Intensive Care Units in 2017 in France: A Nationwide Retrospective Observational Cohort Study Using Data From the French Hospital Discharge Database
Brief Title: Intra Hospital Mortality Risk Factors in Patients Admitted to Cardiac Intensive Care Units in 2017 in France
Acronym: USIC -BNAT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0429
Record Dates: First submitted 2019-01-24; First posted 2019-02-08 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Heart Disease; Acute Coronary Syndrome; Acute Cardiac Failure; Heart Rhythm Disorders; Valve Pathologies
Keywords: Cardiac intensive care unit; Organization; Prognostic score
MeSH Terms: conditions — Heart Diseases; Acute Coronary Syndrome; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective, observational cohort study.

Objectives:

To identify intra hospital mortality risk factors in patients admitted admitted to cardiac intensive care units (CICU). The clinical main endpoint will be the observed percentage of deaths that occured during the year 2017 in french CICU.

To identify the length of stay key determiners of patients admitted in french CICU.

The study will use data from one of the french nationwide healthcare systems database (SNDS) : the national hospital discharge database (PMSI) to be precise.

ELIGIBILITY:
Inclusion criteria:

* Being admitted at least one time in a french CICU in 2017
* Being covered by the mandatory french national health insurance plan in 2017 without discontinuity

Exclusion criteria:

* Being older than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted (at least one time) in a french CICU in 2017
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 1 day
  Observed percentage of deaths that occured during the year 2017 in french CICU

SECONDARY OUTCOMES:
Length of stay at a CICU | 1 year
  Length of stay at a CICU

CONTACTS AND LOCATIONS:
Overall Officials: François Roubille, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC